CLINICAL TRIAL: NCT06069232
Title: Aortic Valve Diseases RISk facTOr assessmenT and Prognosis modeL Construction (ARISTOTLE)
Brief Title: Aortic Valve Diseases RISk facTOr assessmenT and Prognosis modeL Construction
Acronym: ARISTOTLE
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Hospital of Guangdong Medical University (Other); Second Affiliated Hospital of Shantou University Medical College (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Zhongshan People's Hospital, Guangdong, China (Other); Jieyang People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao-dong Zhuang, Professor, Sun Yat-sen University
Other Study IDs: ARISTOTLE Study
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Aortic Valve Disease
Keywords: aortic stenosis; aortic valve insufficiency; risk factor; prediction model
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a multicenter cohort study including patients diagnosed with aortic valve disease during hospitalization, including aortic insufficiency and aortic valve stenosis. The primary outcome of the study was all-cause death, and the secondary outcome was cardiovascular events. Through follow-up observation, the prognostic risk factors of patients with aortic disease were evaluated, and a prognostic model was constructed to guide clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* diagnosed as aortic valve disease

Exclusion Criteria:

* aortic valve replacement at baseline

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participant included in this study were patients with aortic valve disease diagnosed during hospitalization, and these patients were followed up for a long time after discharge.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | from baseline to death or end of follow-up
  death caused by any cause

SECONDARY OUTCOMES:
Cardiovascular death | from baseline to death or end of follow-up
  Death caused by cardiac causes
Aortic valve replacement | from baseline to aortic valve replacement
  Transcatheter aortic valve replacement or surgical aortic valve replacement

CONTACTS AND LOCATIONS:
Overall Officials: xiaodong zhuang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (7):
- China (7):
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sun University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Second Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Eighth Affiliated Hospital, Sun Yat-Sen University, Shenzhen, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong

REFERENCES:
- [Derived] Guo Z, Xiong Z, Zhang W, Chen G, Xie M, Zhou Z, Zhang S, Liu M, Li J, Liao X, Zhuang X. Association between cholesterol, high-density lipoprotein, and glucose index and risks of cardiovascular and all-cause mortality in patients with calcific aortic valve stenosis: the ARISTOTLE cohort study. Cardiovasc Diabetol. 2025 Oct 11;24(1):393. doi: 10.1186/s12933-025-02906-2. PMID 41076530
- [Derived] Li B, Zhang S, Xu C, Huang M, Xiong Z, Hui Z, Liao X, Li J, Chen J, Zhuang X. Association Between the Malnutrition Status and All-Cause Mortality in Patients With Moderate and Severe Aortic Stenosis: A Prospective Cohort Study. J Am Heart Assoc. 2025 Feb 4;14(3):e037086. doi: 10.1161/JAHA.124.037086. Epub 2025 Feb 3. PMID 39895526